CLINICAL TRIAL: NCT01841697
Title: A Phase III, Multicenter, Double-Blind, Randomized Study to Evaluate the Safety and Efficacy of the Addition of MK-3102 Compared With the Addition of Sitagliptin in Subjects With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin
Brief Title: Study to Evaluate the Safety and Efficacy of the Addition of Omarigliptin (MK-3102) Compared With the Addition of Sitagliptin in Participants With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin (MK-3102-026)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3102-026; 2013-000059-42 (EudraCT Number)
Record Dates: First submitted 2013-04-24; First posted 2013-04-26 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Glimepiride; Metformin; Hypoglycemic Agents; Physiological Effects of Drugs; Pharmacologic Actions
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine; Sitagliptin Phosphate; Metformin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omarigliptin 25 mg once weekly (Experimental): Participants receive omarigliptin 25 mg once a week plus placebo to sitagliptin once daily for 24 weeks. Participants continue pre-study stable dose of metformin (total daily dose ≥1500 mg) throughout the study. Participants may receive glimepiride (total daily dose of 1-6 mg) as rescue therapy.
  Interventions: Drug: Omarigliptin; Drug: Placebo to Sitagliptin; Drug: Open-label Metformin; Drug: Open-label Glimepiride
- Sitagliptin 100 mg once daily (Active Comparator): Participants receive sitagliptin 100 mg once daily plus placebo to omarigliptin once a week for 24 weeks. Participants continue pre-study stable dose of metformin (total daily dose ≥1500 mg) throughout the study. Participants may receive glimepiride (total daily dose of 1-6 mg) as rescue therapy.
  Interventions: Drug: Sitagliptin; Drug: Placebo to omarigliptin; Drug: Open-label Metformin; Drug: Open-label Glimepiride

INTERVENTIONS:
Drug: Omarigliptin — Omarigliptin (MK-3102) 25 mg oral capsule once a week for 24 weeks
  Arms: Omarigliptin 25 mg once weekly
Drug: Sitagliptin — Sitagliptin 100 mg oral tablet once a day for 24 weeks
  Arms: Sitagliptin 100 mg once daily
Drug: Placebo to omarigliptin — Placebo to omarigliptin 25 mg oral capsule once a week for 24 weeks
  Arms: Sitagliptin 100 mg once daily
Drug: Placebo to Sitagliptin — Placebo to sitagliptin 100 mg oral tablet once a day for 24 weeks
  Arms: Omarigliptin 25 mg once weekly
Drug: Open-label Metformin — Metformin oral tablet(s) - total daily dose of ≥1500 mg, once or twice a day
  Other Names: Fortamet®; Glucophage®; Glucophage® XR; Glumetza®; Riomet®
Drug: Open-label Glimepiride — Glimepiride oral tablet(s) - total daily dose of 1 to 6 mg once a day as rescue therapy
  Other Names: Amaryl®; Glimy

SUMMARY:
This is a non-inferiority study comparing omarigliptin with sitagliptin in participants with type 2 diabetes mellitus (T2DM) with inadequate glycemic control on metformin therapy. The primary hypothesis is that after 24 weeks, the mean change from baseline in hemoglobin A1c (A1C) in participants treated with omarigliptin is non-inferior to that in participants treated with sitagliptin. There will be a 2-week run-in period with placebo + metformin prior to the double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Currently on a stable dose of metformin monotherapy (≥1500 mg per day) for at least 12 weeks prior to study participation
* Male, or female who is not of reproductive potential or if of reproductive potential agrees to abstain from heterosexual activity or use (or have their partner use) acceptable contraception to prevent pregnancy during the study and for 21 days after the last dose of study drug

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis
* Has been treated with any antihyperglycemic agent (AHA) other than the protocol-required metformin within 12 weeks prior to study participation or with omarigliptin at any time prior to signing informed consent
* History of hypersensitivity to a dipeptidyl peptidase IV (DPP-4) inhibitor
* Is currently participating in, or has participated in, a trial in which the participant received an investigational compound or used an investigational device within the prior 12 weeks of signing the informed consent or is not willing to refrain from participating in any other trial
* History of intolerance, hypersensitivity, or any other contraindication to metformin or sitagliptin
* Is on a weight loss program and is not in the maintenance phase or has been on a weight loss medication in the past 6 months or has undergone bariatric surgery within 12 months prior to study participation
* Has undergone a surgical procedure within 4 weeks of study participation or has planned major surgery during the study
* Is on or likely to require treatment ≥14 consecutive days or repeated courses of corticosteroids (inhaled, nasal and topical corticosteroids are permitted)
* Currently being treated for hyperthyroidism or is on thyroid hormone replacement therapy and has not been on a stable dose for at least 6 weeks
* Is expecting to undergo hormonal therapy in preparation to donate eggs during the period of the trial, including 21 days after the last dose of trial medication
* History of active liver disease (other than non-alcoholic steatosis) including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gall bladder disease
* Human immunodeficiency virus (HIV)
* New or worsening signs or symptoms of coronary heart disease or congestive heart failure within the past 3 months, or myocardial infarction, unstable angina, coronary artery bypass grafting, percutaneous transluminal coronary angioplasty, stroke, or transient ischemic attacks in the past 3 months
* Poorly controlled hypertension
* History of malignancy ≤5 years prior to study participation, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* Hematological disorder (such as aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia)
* Positive urine pregnancy test
* Pregnant or breastfeeding, or is expecting to conceive during the study including 21 days following the last dose of blinded study drug
* User of recreational or illicit drugs or has had a recent history of drug abuse
* Routinely consumes >2 alcoholic drinks per day or >14 alcoholic drinks per week, or engages in binge drinking
* Has donated blood products or has had phlebotomy of >300 mL within 8 weeks of study participation, or intends to donate blood products within the projected duration of the trial or has received, or is anticipated to receive, blood products within 12 weeks of study participation or within the projected duration of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2013-06-13 (Actual); Primary Completion 2014-11-17 (Actual); Study Completion 2014-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Goldenberg R, Gantz I, Andryuk PJ, O'Neill EA, Kaufman KD, Lai E, Wang YN, Suryawanshi S, Engel SS. Randomized clinical trial comparing the efficacy and safety of treatment with the once-weekly dipeptidyl peptidase-4 (DPP-4) inhibitor omarigliptin or the once-daily DPP-4 inhibitor sitagliptin in patients with type 2 diabetes inadequately controlled on metformin monotherapy. Diabetes Obes Metab. 2017 Mar;19(3):394-400. doi: 10.1111/dom.12832. Epub 2017 Jan 17. PMID 28093853
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=3102-026&kw=3102-026&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Omarigliptin 25 mg Once Weekly: Participants received omarigliptin 25 mg once a week plus placebo to sitagliptin once daily for 24 weeks. Participants continued pre-study stable dose of metformin (total daily dose ≥1500 mg) throughout the study. Participants may have received glimepiride (total daily dose of 1-6 mg) as rescue therapy.
- Sitagliptin 100 mg Once Daily: Participants received sitagliptin 100 mg once daily plus placebo to omarigliptin once a week for 24 weeks. Participants continued pre-study stable dose of metformin (total daily dose ≥1500 mg) throughout the study. Participants may have received glimepiride (total daily dose of 1-6 mg) as rescue therapy.
Period: Overall Study
Arm/Group | Omarigliptin 25 mg Once Weekly | Sitagliptin 100 mg Once Daily
Started | 322 | 320
Completed | 302 | 302
Not Completed | 20 | 18
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 16 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omarigliptin 25 mg Once Weekly | Sitagliptin 100 mg Once Daily | Total
Number analyzed (Participants) | 322 | 320 | 642
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.0 (9.8) | 57.6 (9.8) | 57.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 145 | 316
  Male | 151 | 175 | 326
Hemoglobin A1c (A1C) [Mean (Standard Deviation); unit: Percent] | 7.52 (0.77) | 7.49 (0.74) | 7.50 (0.76)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 160.1 (35.7) | 153.9 (32.8) | 157.0 (34.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at Week 24
Description: A1C is a measure of the percentage of glycated hemoglobin in the blood. Participant whole blood samples were collected at baseline and Week 24 to determine the least squares mean A1C change from baseline.
Time Frame: Baseline and Week 24
Population: Full analysis set population consists of all randomized participants who received at least one dose of study treatment and have a baseline measurement or a post-randomization measurement for the analysis endpoint subsequent to at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Omarigliptin 25 mg Once Weekly | Sitagliptin 100 mg Once Daily
Number analyzed (Participants) | 322 | 320
Percent | -0.47 [-0.55 to -0.38] | -0.43 [-0.51 to -0.35]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg Once Weekly vs Sitagliptin 100 mg Once Daily; Constrained longitudinal data analysis; Test type: Non-Inferiority or Equivalence — If the upper bound of the two-sided 95% confidence interval for the mean difference between omarigilptin and sitagliptin is less than the non-inferiority margin, δ =0.3%, then omarigliptin will be declared non-inferior to sitagliptin in terms of A1C reduction at Week 24; Difference in least squares mean = -0.03, 95% CI 2-sided [-0.15 to 0.08] — Difference is omarigliptin minus sitagliptin

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event
Description: An adverse event is defined as any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event. Data presented below excludes data after initiation of glycemic rescue therapy.
Time Frame: Up to 27 weeks (including 3-week follow-up)
Population: All participants as treated population consists of all randomized participants who received at least one dose of trial treatment. Participants are included in the treatment group corresponding to the trial treatment they actually received.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin 25 mg Once Weekly | Sitagliptin 100 mg Once Daily
Number analyzed (Participants) | 322 | 320
Percentage of participants | 36.3 | 40.6
Statistical Analysis 1: Comparison: Omarigliptin 25 mg Once Weekly vs Sitagliptin 100 mg Once Daily; Test type: Superiority or Other; Difference in percent = -4.3, 95% CI 2-sided [-11.8 to 3.2] — Difference is omarigliptin minus sitagliptin

3. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: as for outcome 2
Time Frame: Up to 24 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin 25 mg Once Weekly | Sitagliptin 100 mg Once Daily
Number analyzed (Participants) | 322 | 320
Percentage of participants | 0.9 | 2.2
Statistical Analysis 1: Comparison: Omarigliptin 25 mg Once Weekly vs Sitagliptin 100 mg Once Daily; Test type: Superiority or Other; Difference in percent = -1.3, 95% CI 2-sided [-3.6 to 0.8] — Difference is omarigliptin minus sitagliptin

4. Secondary Outcome: Change From Baseline in FPG at Week 24
Description: Participant whole blood samples were collected after an overnight fast at baseline and Week 24 to determine the least squares mean change from baseline in participant FPG.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin 25 mg Once Weekly | Sitagliptin 100 mg Once Daily
Number analyzed (Participants) | 322 | 320
mg/dL | -13.7 [-17.3 to -10.1] | -9.5 [-13.2 to -5.9]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg Once Weekly vs Sitagliptin 100 mg Once Daily; Test type: Superiority or Other; p = 0.089, Constrained logitudinal data analysis; Terms for treatment, time, and the interaction of time by treatment, with the constraint that the mean baseline is the same for all treatment groups; Difference in least squares mean = -4.2, 95% CI 2-sided [-9.0 to 0.6] — Difference is omarigliptin minus sitagliptin

5. Secondary Outcome: Percentage of Participants Achieving an A1C Goal <7.0% After 24 Weeks of Treatment
Description: Participant whole blood samples were collected at Week 24 to determine the number of participants achieving A1C <7.0% at Week 24.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin 25 mg Once Weekly | Sitagliptin 100 mg Once Daily
Number analyzed (Participants) | 322 | 320
Percentage of participants | 50.9 [48.8 to 59.9] | 49.1 [46.8 to 57.9]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg Once Weekly vs Sitagliptin 100 mg Once Daily; Proportion (rate) for each group was estimated using standard multiple imputation techniques. Between-group difference in proportion is omarigliptin minus sitagliptin; Test type: Superiority or Other; p = 0.619, Miettinen & Nurminen method; Between-group rate difference = 2.0, 95% CI 2-sided [-5.9 to 9.9]

6. Secondary Outcome: Percentage of Participants Achieving an A1C Goal <6.5% After 24 Weeks of Treatment
Description: Participant whole blood samples were collected at Week 24 to determine the percentage of participants achieving A1C <6.5% at Week 24.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin 25 mg Once Weekly | Sitagliptin 100 mg Once Daily
Number analyzed (Participants) | 322 | 320
Percentage of participants | 27.0 [24.0 to 34.1] | 22.8 [19.9 to 29.5]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg Once Weekly vs Sitagliptin 100 mg Once Daily; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.212, Miettinen & Nurminen method; Between-group rate difference = 4.4, 95% CI 2-sided [-2.5 to 11.4]

ADVERSE EVENTS:
Time Frame: Up to 27 weeks (including 3-week follow-up)
Description: All participants as treated population defined as all randomized participants who received at least 1 dose of study drug. Participants are included in the treatment group corresponding to the trial treatment they actually received. Serious and non-serious AEs, respectively, include and exclude data after the initiation of glycemic rescue therapy.
Arm/Group | Omarigliptin 25 mg Once Weekly | Sitagliptin 100 mg Once Daily
Serious Adverse Events (participants affected / at risk) | 11/322 | 9/320
Other Adverse Events (participants affected / at risk) | 0/322 | 0/320
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin 25 mg Once Weekly (N=322) | Sitagliptin 100 mg Once Daily (N=320)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Sebaceous adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dematitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.